CLINICAL TRIAL: NCT04517474
Title: Evaluación de Una Herramienta E-Salud Para la reducción Del Consumo de Cannabis
Brief Title: Comparing the Spanish Version of CANreduce With or Without Psychological Support and Treatment as Usual, Reducing Cannabis Use.
Acronym: CANREDUCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Research Institute for Public Health and Addiction, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/8901/I
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Cannabis Use Disorder
Keywords: Mental health; Adherence, Treatment; Cognitive behavioral therapy; Web-based Self-Help
MeSH Terms: conditions — Psychological Well-Being; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Masking Description: The masking technique will be partially single-blinded-in that participants in either of the two active treatment groups will not know which version they work with. The two versions are neutrally described as two differently optimized variants to prevent participants from having a preference of one over the other possibly resulting in a disappointment when being allocated to the unwished version. However, subjects will know whether they have been assigned to treatment-as-usual (TAU). Any blinding of research and study personnel is not warranted.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CANreduce with psychological support (Experimental): Adherence-focused guidance enhanced web-based self-help for the reduction of cannabis use with psychological support
  Interventions: Behavioral: CANreduce; Behavioral: psychological support
- CANreduce without psychological support (Experimental): Adherence-focused guidance enhanced web-based self-help for the reduction of cannabis use without psychological support
  Interventions: Behavioral: CANreduce
- Treatment as usual (No Intervention): Users will be prompt to a web with a list of the treatment centers nearby their postal code

INTERVENTIONS:
Behavioral: CANreduce — CANreduce is an automated web-based self-help tool based on classical Cognitive Behavioral Treatment (CBT) approaches for treating cannabis dependence. It will consist of a consumption diary, eight modules designed to reduce cannabis use based on the principles of motivational interviewing, self-control practices, and methods of cognitive behavioral therapy ( strategies for goal achievement, Identifying risk situations, Dealing with cannabis craving, Dealing with relapses, Working on needs, Saying "no" to foster refusal skills, Dealing with burdens, Preserving achievements). Participants can study all modules at their own pace and order, though a specific order will be advised.
  Other Names: CANreduce: Adherence-focused guidance enhanced web-based self-help for the reduction of cannabis use with psychological support
  Arms: CANreduce with psychological support; CANreduce without psychological support
Behavioral: psychological support — psychological support
  Arms: CANreduce with psychological support

SUMMARY:
Cannabis is the most widely used psychoactive substance around the world after alcohol and tobacco. Although approximately one in ten users develop serious problems of dependency, only a small number attend outpatient addiction counseling centers. CANreduce is an adherence-focused guidance enhanced web-based self-help program with promising results in German and other languages. It also reaches those users who hesitate to approach such treatment centers and help them to reduce their cannabis use.

This study will test the effectiveness of the Spanish version of the enhanced web-based self-help intervention with psychological support, an enhanced web-based self-help intervention (without psychological support) and a waiting list control in reducing cannabis use in problematic users.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis use of at least once a week 30 days prior to study entry
* At least 18 years old
* At least weekly internet access and a valid email address

Exclusion Criteria:

* Participant reports current pharmacological psychiatric disease or history of psychosis, schizophrenia, bipolar type I disorder or significant current suicidal or homicidal thoughts
* Use of other pharmacological and psychosocial treatments for cannabis use disorders
* Inability to read or write in Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of days of self-reported cannabis use in the past 30 days (TLFB) | Baseline, 6, 12 and 24 weeks.
  Participants enter their cannabis consumption frequency into their consumption diary every week.
  More days of self-reported cannabis use indicate worse state

SECONDARY OUTCOMES:
Change in the number of days of weekly self-reported cannabis use Time Life Follow Back (TLFB) | Baseline, 6, 12 and 24 weeks.
  Participants enter their cannabis consumption frequency into their consumption diary every week.
  More days of self-reported cannabis use indicate a worse outcome
Change in the quantity of weekly standard joints (TLFB with predifined cannabis standard joints) | Baseline, 6, 12 and 24 weeks.
  Participants enter their cannabis consumption quantity into their consumption diary every week.
  More number of weekly standard joints indicate a worse outcome
Change in the scoring of the Cannabis Use Disorder Identification Test - Revised (CUDIT-R) | Baseline, 6, 12 and 24 weeks.
  CUDIT-R was developed containing 8 items, two each from the domains of consumption, cannabis problems (abuse), dependence, and psychological features. It has excellent psychometric properties. High sensitivity (91%) and specificity (90%).
  This questionnaire was designed for self administration and is scored by adding each of the 8 items:
  * Question 1-7 are scored on a 0-4 scale (range 0-28)
  * Question 8 is scored 0, 2 or 4.
  * Score range 0-32 Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder for which further intervention may be required.
  Higher scores indicate a worse outcome
Change in the scoring of the Severity Dependence Scale (SDS) | Baseline, 6, 12 and 24 weeks.
  SDS is a standard instrument to assess the severity to any drug dependence. Each of the five items is scored on a 4-point scale (0-3). The total score is obtained through the addition of the 5-item ratings (0-15). The higher the score the higher the level of dependence.
Change in the scoring of the Alcohol Use Disorders Identification Test (AUDIT) | Baseline, 6, 12 and 24 weeks.
  AUDIT is a 10-item screening tool developed by the World Health Organization (WHO) to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Each item scores 0-4, The total score ranges from 0-40. A score of 8 or more is considered to indicate hazardous or harmful alcohol use. The AUDIT has been validated across genders and in a wide range of racial/ethnic groups and is well suited for use in primary care settings. Higher scores indicate a worse outcome
Change in the scoring of the PROMIS Emotional Distress - Depression - Short Form 8b | Baseline, 6, 12 and 24 weeks.
  PROMIS (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Developed and validated with state-of-the-science methods to be psychometrically sound and to transform how life domains are measured.
  8 items 1-5, score ranges 8-40 Higher scores indicate a worse outcome
Change in the scoring of the PROMIS Anxiety 8a - Adult v1.0 | Baseline, 6, 12 and 24 weeks.
  PROMIS (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. Developed and validated with state-of-the-science methods to be psychometrically sound and to transform how life domains are measured.
  8 items 1-5, score ranges 8-40 Higher scores indicate a worse outcome
Change in the scoring of the EQ-5D-5L | Baseline, 6, 12 and 24 weeks.
  EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Score ranges from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health),
  The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Torrens, PhD, Principal Investigator — Hospital del Mar Research Institute (IMIM)
Locations (1):
- Juan-Ignacio Mestre-Pinto, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amann M, Haug S, Wenger A, Baumgartner C, Ebert DD, Berger T, Stark L, Walter M, Schaub MP. The Effects of Social Presence on Adherence-Focused Guidance in Problematic Cannabis Users: Protocol for the CANreduce 2.0 Randomized Controlled Trial. JMIR Res Protoc. 2018 Jan 31;7(1):e30. doi: 10.2196/resprot.9484. PMID 29386176
- [Background] Schaub MP, Wenger A, Berg O, Beck T, Stark L, Buehler E, Haug S. A Web-Based Self-Help Intervention With and Without Chat Counseling to Reduce Cannabis Use in Problematic Cannabis Users: Three-Arm Randomized Controlled Trial. J Med Internet Res. 2015 Oct 13;17(10):e232. doi: 10.2196/jmir.4860. PMID 26462848
- [Derived] Mestre-Pinto JI, Fonseca F, Schaub MP, Baumgartner C, Alias-Ferri M, Torrens M. CANreduce-SP-adding psychological support to web-based adherence-focused guided self-help for cannabis users: study protocol for a three-arm randomized control trial. Trials. 2022 Jun 22;23(1):524. doi: 10.1186/s13063-022-06399-2. PMID 35733201
- See also: Web of the Spanish study (in Spanish) — http://canreduce.es
- See also: Web of the Swiss study (in German) — http://canreduce.at